CLINICAL TRIAL: NCT00455559
Title: A Phase II Study of Perifosine Plus Imatinib Mesylate for Patients With Resistant Gastrointestinal Stromal Tumor
Brief Title: Ph II Study of Perifosine Plus Gleevec for Patients With GIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 210
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2011-11

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Resistant Gastrointestinal Stromal Tumor; GIST; Perifosine; Gleevec
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — perifosine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perifosine 100 mg/d + imatinib mesylate (Experimental): Perifosine 100 mg/d x 28 days Oral daily dose of perifosine 100 mg and oral daily dose of imatinib mesylate (current dose at time of progression of disease [PD] without interruption). Both drugs will be taken on a continuous basis and should be taken with food. Each cycle will be defined as 28 days.
  Interventions: Drug: Perifosine; Drug: Imatinib Mesylate
- Perifosine 900 mg/d + imatinib mesylate (Experimental): Perifosine 900 mg/d (300 mg tid), 1 x weekly Oral once-weekly dose of perifosine 900 mg (300 mg tid) + oral daily dose of imatinib mesylate (current dose at time of PD without interruption). Perifosine will be taken on days 1, 8, 15, and 22 of a 28-day cycle. Both medications should be taken with food.
  Interventions: Drug: Perifosine; Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Perifosine
  Other Names: D-21266; KRX-0401
Drug: Imatinib Mesylate
  Other Names: Gleevec; STI-571

SUMMARY:
This is a Phase II trial designed to determine the efficacy and safety of perifosine plus imatinib mesylate in patients with advanced GIST who develop progressive disease or recurrence while receiving imatinib mesylate.

DETAILED DESCRIPTION:
This is a Phase II study of perifosine in combination with imatinib mesylate in patients with advanced GIST. Each cycle lasts 28 days. There will be two treatment arms. On both arms, patients will continue the dose of imatinib mesylate taken during the period of disease progression. Patients will be randomized to one either a weekly or a daily perifosine treatment regimen at the time of registration.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed diagnosis of Kit expressing advanced GIST. This includes patients with metastatic disease or with primary tumors that are considered inoperable.
* Patients may have "limited" (some but not all tumor foci progressing that are not amenable to local therapy) or "generalized" (widespread growth of all tumor foci) progression after adequate therapy with imatinib mesylate. Patients must have progression of disease on imatinib mesylate (at any dose greater than or equal to 300 milligrams daily).
* Patients must have documented measurable disease by CT scan (> 2 cm by conventional CT or > 1 cm by spiral CT). If a targeted lesion has been previously embolized or irradiated, there must be objective evidence of progression of the lesion per CT scan, post-embolization or in the radiated field.
* Patients must be at least four weeks out and recovered from acute toxicities of prior therapy, including radiation, biotherapy, chemotherapy or embolization (with the exception of imatinib mesylate).
* All patients must have progressive disease on imatinib defined as:

  * An increase in unidimensional tumor size of >10% and did not meet criteria for PR by CT density
  * Any new lesions, including new tumor nodules in a previously cystic tumor, while on imatinib therapy
* Patients should have a performance status of 0 to 2 according to the ECOG criteria.
* Patients must have adequate organ function, unless in the opinion of the treating investigator, the abnormality is related to tumor and the study chairman or medical monitor agree the abnormality is unlikely to affect the safety of perifosine use. Adequate organ and marrow function is described in the protocol.
* Patients must be able to ingest oral medications or to obtain them through a gastrostomy tube.
* Patients must have ability to understand and the willingness to sign a written informed consent document.
* Patients must be at least 18 years of age

Exclusion Criteria

* Presence of known symptomatic CNS metastases
* Significant concurrent medical disease other than GIST, including:

  * New York Heart Association class III or IV cardiac problems (e.g., congestive heart failure, acute myocardial infarction within 2 months of study), uncontrolled chronic renal
  * liver disease
  * uncontrolled diabetes
  * uncontrolled seizure disorder
  * active uncontrolled infection
  * organ allografts
  * psychiatric illness/social situations that would limit compliance with study requirements
* History of active secondary cancer, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 or more years.
* Patients who are receiving any other investigational agents or devices.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine.
* Female patients who are pregnant or lactating are ineligible. All females of childbearing potential must have a negative serum pregnancy test within 72 hours of treatment. Men and women of childbearing potential must agree to employ adequate contraception to prevent pregnancy while on therapy and for 4 weeks after the completion of treatment. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy and safety of perifosine plus imatinib mesylate in patients with advanced GIST who develop progressive disease or recurrence while receiving imatinib mesylate. | Every 8 weeks
  This is a two-arm Phase II trial to determine whether the experimental regimen is likely to provide a 20% response rate while controlling the toxicity rate at 15%. Response will be evaluated at 2 months from the start of therapy, and is defined using the Choi Criteria. Toxicity is defined as any of the following events: regimen-related death, grade 3 transaminitis, grade 3 gastrointestinal toxicity, or grade 4 fatigue or higher within the same 2-month time window.

SECONDARY OUTCOMES:
To determine whether inhibition of Akt phosphorylation correlates with survival, time to disease progression, or response rate in patients with advanced GIST treated with imatinib mesylate plus perifosine. | Every 8 weeks
  As perifosine inhibits activation of Akt and has an acceptable safety profile, this Phase II trial is designed to assess antitumor activity of perifosine in patients with advanced GIST who are refractory to or relapsed from imatinib mesylate.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Trent, MD, PhD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- [Result] Journal of Clinical Oncology, 2009 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 27, No 15S (May 20 Supplement), 2009: 10563